CLINICAL TRIAL: NCT00771732
Title: Noveon Laser Treatment of Onychomycosis: A Device Performance Clinical Study
Brief Title: Using Light Therapy to Treat Toe Nail Fungus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nomir Medical Technologies (Industry)
Responsible Party: Nomir Medical Technologies, Nomir Medical Technologies
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 09.002; 07-301
Record Dates: First submitted 2008-07-07; First posted 2008-10-13 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Onychomycosis
Keywords: toe nail fungus
MeSH Terms: conditions — Onychomycosis | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Light therapy
  Interventions: Device: light therapy
- 2 (Sham Comparator): 6 minute "session" given with machine "off"
  Interventions: Device: light therapy

INTERVENTIONS:
Device: light therapy — 6 minute light therapy
  Other Names: laser threapy
  Arms: 1
Device: light therapy — combination of wavelengths
  Other Names: No therapy/machine is "off"
  Arms: 2

SUMMARY:
To see if four sessions of light therapy successfully treats nail fungus.

DETAILED DESCRIPTION:
This study is a one year study which includes four treatment sessions of light therapy looking for clinical and mycological improvement.

ELIGIBILITY:
Inclusion Criteria:

* toe nail fungus, not infolving lunula
* between ages 18-70 years old

Exclusion Criteria:

* not on systemic anti-fungal medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
clinical improvement | six months

SECONDARY OUTCOMES:
mycological negative | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Robbins, M.D., Study Chair — Nomir Medical Technologies
Locations (1):
- Paula Angelini, DPM, Southborough, Massachusetts, United States